CLINICAL TRIAL: NCT00101881
Title: Transthoracic Incremental Monophasic Versus Biphasic by Emergency Responders (TIMBER)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Medic One Foundation (Other)
Responsible Party: Peter J. Kudenchuk, MD, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00-3776-B05
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-09

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Defibrillation; Biphasic defibrillation; Monophasic defibrillation; Ventricular fibrillation
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monophasic Shock (Active Comparator): Administration of monophasic waveform defibrillation
  Interventions: Device: Defibrillation (biphasic versus monophasic shock)
- Biphasic Shock (Active Comparator): Administration of biphasic waveform defibrillation
  Interventions: Device: Defibrillation (biphasic versus monophasic shock)

INTERVENTIONS:
Device: Defibrillation (biphasic versus monophasic shock) — Administration of monophasic or biphasic waveform defibrillation

SUMMARY:
The study compares the effectiveness of two fully approved shock waveforms (monophasic and biphasic shock) commonly used to defibrillate (shock) patients with out-of-hospital cardiac arrest due to a highly lethal rhythm problem (ventricular fibrillation). The purpose of the study (hypothesis) is to determine if one waveform results in improved resuscitation, admission alive to hospital, and discharge alive from hospital compared with the other.

DETAILED DESCRIPTION:
The trial is designed to determine whether two fully-FDA-approved, commercially available transthoracic defibrillation shock waveforms at comparable energies result in improved patient outcome following out-of-hospital cardiac arrest due to ventricular fibrillation. Eligible subjects include all adults with nontraumatic out-of-hospital cardiac arrest due to ventricular fibrillation. Subjects in cardiac arrest will be randomly allocated to receive one of two types of defibrillation shocks (monophasic or biphasic waveform) during their resuscitation, which will in addition include all other standard treatments. The primary endpoint is admission alive to hospital. Secondary endpoints include rhythm after defibrillation shock, return of spontaneous circulation, and hospital discharge rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult victims of nontraumatic out-of-hospital cardiac arrest due to ventricular fibrillation

Exclusion Criteria:

* Children
* Trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2002-11; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Admission alive to hospital | Within hours of intervention

SECONDARY OUTCOMES:
Rhythm after defibrillation shock | Within minutes of intervention
Return of spontaneous circulation | Within minutes of intervention
Hospital discharge rates | Within days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Kudenchuk, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Kudenchuk PJ, Cobb LA, Copass MK, Olsufka M, Maynard C, Nichol G. Transthoracic incremental monophasic versus biphasic defibrillation by emergency responders (TIMBER): a randomized comparison of monophasic with biphasic waveform ascending energy defibrillation for the resuscitation of out-of-hospital cardiac arrest due to ventricular fibrillation. Circulation. 2006 Nov 7;114(19):2010-8. doi: 10.1161/CIRCULATIONAHA.106.636506. Epub 2006 Oct 23. PMID 17060379